CLINICAL TRIAL: NCT04571268
Title: Motions of the Bones and Activation of the Muscles of the Shoulder Girdle During Basic and Common Arm Movement
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: More Foundation (Other)
Collaborators: DePuy Synthes Products, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 4030
Record Dates: First submitted 2020-09-12; First posted 2020-10-01 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-10

CONDITIONS: Rotator Cuff Tears
Keywords: Rotator cuff tear; Shoulder motion; Shoulder muscle activation
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy validation subjects: Healthy subjects who meet the inclusion criteria and participate in data collection for the purpose of developing and validating the biomechanical models used to track scapular motion
- Healthy comparison subjects: Healthy subjects who meet the inclusion criteria and participate in data collection for comparison of shoulder motion and muscle activation patterns with RCT subjects
- RCT subjects: Subjects who have sustained a major rotator cuff tear

SUMMARY:
A comprehensive understanding of healthy shoulder motion is a valuable contribution to the academic literature and provides a basis of comparison for various shoulder pathologies and treatments. However, the medical community is primarily interested in how pathology affects shoulder function and the underlying musculoskeletal reasons for impaired function associated with specific pathologies. Rotator cuff tears (RCT) provide an excellent model to study shoulder biomechanics because RCTs can cause significant functional impairment and can be quantified in size and location using standard clinical imaging techniques.

Upon completion of this study a comprehensive database of three-dimensional joint angles and EMG patterns of the structures of the shoulder joint complex of dominant and non-dominant during common activities of daily living will be available for healthy subjects and those of subjects whose dominant limbs are impaired by rotator cuff tears. These data will show normal muscle activations and movement patterns required to complete activities of daily living and compare them to the movement, and muscle activation patterns of persons who exhibit muscular and movement dysfunction due to rotator cuff tears.

DETAILED DESCRIPTION:
Rotator cuff tears occur in approximately 20% of patients older than 65 years and increase with age. These non-traumatic RCTs are generally caused by normal age-related degeneration. Surgical treatment is effective, however recurrence of injury is common especially when the original tear was caused by age related degeneration. Non-surgical treatment options are designed to decrease pain and improve performance of activities of daily living and may be an effective alternative to surgery. If non-surgical treatment options are unsuccessful, surgical treatment may be considered. When rotator cuff tears are treated surgically, postoperative rehabilitation is an important factor in determining outcome success, however there is uncertainty regarding the best protocols for post-surgery rehabilitation. Evidence suggests that a more complete understanding of motion and muscle activation is necessary to design effective and reliable rehabilitation programs for rotator cuff injuries.

These data will enable medical professionals to better answer a range of clinical questions. They will provide health care professionals and researchers with a knowledge of relative muscle contributions to specific joint motions required to perform activities of daily living. This information is well suited to refine input variables for computer models and robotic testing platforms which can improve virtual and cadaver testing of shoulder impairment and repair models. Understanding the limitations to movement caused by RCT, and the resulting muscle activation patterns, will inform better surgical indications and enable therapists to better design rehabilitation protocols to enhance recovery from rotator cuff tears with or without surgery, as well as develop programs to limit future tears. Knowledge of muscle activation patterns during activities of daily living will also allow pre-habilitation protocols to be tailored for a subsequent surgical procedure such as reverse shoulder arthroplasty. These data will also assist in the design of shoulder prostheses whose biomechanical characteristics will compensate for deficiencies present in a shoulder joint impaired by rotator cuff injury. The knowledge gained from this study will provide a basis for future studies investigating traumatic shoulder injuries and the design of effective rehabilitation protocols for such injuries.

ELIGIBILITY:
Inclusion Criteria:

All subjects

* Right hand dominant
* English speaking
* Subjects who have read and signed IRB approved informed consent for the study.

RCT subjects:

* Chronic right-side side shoulder pain with documented rotator cuff tear involving 2 or more tendons, and greater than 5cm as diagnosed by MRI
* Exhibit right rotator cuff disfunction without corresponding changes in the glenohumeral joint.
* Weakness of right rotator cuff isolated function based on clinical exam findings.
* Fatty infiltration grade 2 or more for involved muscle bellies based on MRI findings.

Exclusion Criteria:

* Unable to achieve 30º of external rotation and 140º of elevation in the scapular plane, where the limitations are not due to cuff tear associated pain.
* Diagnosis of osteoarthritis of the shoulder on their right side.
* History of musculoskeletal injury or disorder affecting any part of the right arm except the rotator cuff of the shoulder.
* History of musculoskeletal injury or disorder affecting any part of the left arm.
* Any musculoskeletal injury or disorder which prevents the subject standing unassisted for an extended period.
* Parkinson's disease.
* History of cerebral vascular accident.
* Pregnant.
* Current Incarceration.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients between 50 and 70 years old, inclusive, who present with chronic right shoulder pain with a documented right rotator cuff tear will be screened for eligibility and participation. Rotator cuff tear subjects will be recruited under consultation with physicians from their patient populations. Patient charts will be assessed by study investigators to ensure they meet inclusion/exclusion criteria prior to consent. Healthy subjects will be recruited by flyer and word of mouth from the surrounding general population. Healthy subjects will be of similar demographics to the rotator cuff tear subjects.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-01-28 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Range of motion | At enrollment
  Measure range of motion in abduction, forward flexion, external rotation in neutral position and external rotation at 90 degrees abductions with corresponding rotator cuff muscle activation patterns
Activities of Daily Living | At enrollment
  Measure glenohumeral joint angles and rotator cuff muscle activation patterns during the performance of prescribed activities of daily living

SECONDARY OUTCOMES:
Patient reported outcome | At enrollment
  Completion of QuickDASH questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Marc D Jacofsky, PhD, Study Director — More Foundation
Locations (1):
- MORE Foundation, Phoenix, Arizona, United States